CLINICAL TRIAL: NCT01499823
Title: Permeability Map As an Imaging Biomarker to Distinguish Progression From Pseudoprogression in High-Grade Glioma
Brief Title: Permeability Map to Distinguish Progression From Pseudoprogression in High-Grade Glioma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Hong Choi, Seoul National University Hospital, Seoul National University Hospital
Other Study IDs: H-1108-032-372
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: High Grade Glioma
Keywords: Permeability Map; High-Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with high-grade glioma: Patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who receive concurrent chemoradiation (CCRT) with temozolomide

SUMMARY:
The aim of the present study is to assess whether a new method of quantifying therapy-associated hemodynamic alterations based on DCE MR imaging may help to distinguish pseudoprogression from true progression in patients with high grade glioma, who received CCRT.

DETAILED DESCRIPTION:
Combination temozolomide and radiation significantly prolongs survival compared with radiation alone and has become standard treatment for glioblastoma multiforme (GBM). Response assessment in GBM is difficult as a result of the frequent occurrence of early imaging changes indistinguishable from tumor progression, termed pseudoprogression. The majority of patients remain clinically stable. It is often unclear whether current therapy should be maintained or second-line therapy initiated. The incidence of pseudoprogression after concurrent chemoradiation is15%to 30%. A potential mechanism of pseudoprogression is that radiation-induced vascular changes may lead to focal transient increase in gadolinium enhancement. Dynamic contrast-enhanced (DCE) MR imaging provides a noninvasive means for quantifying tumor vascular properties.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who received concurrent chemoradiation (CCRT) with temozolomide, the patients show the measurable enhancing portion (1 cm in the long diameter according to the RANO criteria) in the immediate f/up MRI after CCRT.

Exclusion Criteria:

* Among the patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who received concurrent chemoradiation (CCRT) with temozolomide, the patients do not show the measurable enhancing portion (1 cm in the long diameter according to the RANO criteria) in the immediate f/up MRI after CCRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma), who receive concurrent chemoradiation (CCRT) with temozolomide
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Permeability Map to Distinguish Progression From Pseudoprogression in High-grade glioma | 2year

CONTACTS AND LOCATIONS:
Overall Officials: SeungHong Choi, MD, PhD, Principal Investigator — Seoul National University Hospital(Radiology)
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea